CLINICAL TRIAL: NCT06365567
Title: Evaluation of Liver and Osteo-metabolic Complications Related to the Consumption of Fructose in a Cohort of Overweight and Obese Children and Adolescents.
Brief Title: Dietary Fructose: a Metabolic Switch in Pediatric Obesity-related Disease.
Acronym: EO2022
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Collaborators: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Responsible Party: Principal Investigator, Flavia Prodam, Professor, Azienda Ospedaliero Universitaria Maggiore della Carita
Other Study IDs: CE209/2023
Record Dates: First submitted 2024-02-12; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Pediatric Obesity
Keywords: pediatric; obesity; NAFLD; Fructose
MeSH Terms: conditions — Pediatric Obesity; Obesity; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The increase in childhood obesity is a multifactorial phenomenon influenced by dietary patterns, commercial factors, and social determinants; it has long-term consequences for both individual health and society as a whole. Despite recommendations for maintaining good health throughout life and promoting the Mediterranean Diet, due to the increased availability of ultra-processed and more appealing foods, children and adolescents are shifting towards a "Western" diet. One in four children consumes sugary and carbonated drinks every day, which contributes to a high intake of fructose in the diet, while fruits and vegetables are consumed less, and legumes are included in the diet of only 38% of children less than once a week.

Fructose is a monosaccharide naturally found in fruits, vegetables, and honey; due to its high sweetness and taste-enhancing properties, fructose is widely used in the food industry. High-fructose corn syrup, in particular, is one of the most widely used ingredients in the production of soft drinks, jams, breakfast cereals, and bakery products. Non-alcoholic fatty liver disease (NAFLD), now also called metabolic dysfunction-associated fatty liver disease (MAFLD), is considered the hepatic manifestation of metabolic syndrome and currently represents the most common chronic liver disease in pediatric age in Western countries. Recent studies suggest that fructose consumption is implicated in the development of NAFLD both directly by providing metabolites that can be used for triglyceride and free fatty acid synthesis, and indirectly through increased uric acid production. High-fructose foods also appear to be a risk factor for bone loss. Numerous studies conducted over the past 25 years, during which fructose consumption has exponentially increased, have shown that this sweetener tends to increase the incidence of fractures and osteoarthritis and decrease bone mineral density (BMD) and new bone tissue deposition.

The objective of this study is to understand the effect of fructose on the molecular events that contribute to the evolution of the pediatric age, and its effective relationship with the onset of liver and osteoarticular complications in this population. Understanding the mechanisms of fructose regulation and its effects on the body could be an important target to address the clinical and social problems arising from its spread in children.

DETAILED DESCRIPTION:
At the time of recruitment, patients referred to the Endocrinology Outpatient Clinic of the AOU (Azienda Ospedaliera Universitaria) Maggiore della Carità in Novara, the Transition Endocrinology Outpatient Clinic of the Endocrinology SCDU (Struttura Complessa a Direzione Universitaria), and the Pediatric Endocrinology Outpatient Clinic "B. Trambusti" of the Giovanni XXIII Pediatric Hospital, will undergo:

Questionnaires to assess the quantity of fructose intake through diet:

* KIDMED (quality index for children and adolescents) questionnaire to evaluate adherence to the Mediterranean diet in children/adolescents.
* IDEFICS (Identification and preven- tion of Dietary- and lifestyle- induced health EFfects In Children and infantS) questionnaire to assess food frequency in children.
* 24-hour recall questionnaire to gather information about meals consumed in the previous 24 hours. Macronutrient quantities will be obtained using dedicated software, "Professional Diet Therapy Software Dietosystem" from DSMedica(industry supplying the software). The questionnaire includes specific questions and figures to identify food portions and relate them to the quantity of fructose consumed.
* Calculation of the Dietary Inflammatory Index (DII) through a list of foods. This parameter allows for the determination of how much a dietary pattern promotes the synthesis of pro-inflammatory molecules.
* Sociological questionnaire prepared ad hoc by Unit 3 to assess dietary habits and fructose intake in relation to the family's socioeconomic status.

Anamnestic evaluation:

* The mother of the patient will be asked for gestational age, mode of delivery, and the child's birth anthropometric data.
* Recording of current pharmacological therapy (if present).

Instrumental evaluation:

* Quantitative and qualitative analysis of bone composition using quantitative ultrasound (QUS). This tool provides various parameters related to bone composition, specifically speed of sound (SOS) for bone density evaluation, broadband ultrasound attenuation (BUA) for trabecular structure evaluation, ultrasound peak amplitude for trabecular size evaluation, number of peaks for connectivity evaluation of the mineralized matrix structure, and energy and amplitude of fast waves for elasticity evaluation.
* Abdominal ultrasound (US) to assess hepatic steatosis, perivisceral and subcutaneous fat. The presence of hepatic steatosis (NAFLD) will be classified from stage 1 to stage 3 according to the literature.

Clinical-auxological evaluation:

* Anthropometric measurements including weight, height, and BMI according to STANDARD DEVIATION SCORE (SDS).
* Waist and hip circumference measurements.
* Measurement of blood pressure and heart rate.
* Analysis of body composition through bioimpedance analysis (BIA).

Expected results With this study, the investigators expect to acquire new knowledge about the effect of fructose on the onset of obesity-associated liver disease (NAFLD) and bone metabolism, by identifying new biological, immunological, and omics markers that can be studied in the future as disease targets in the pediatric population. Furthermore, due to scientific and sociological interest, this study aims to identify sociodemographic and cultural determinants related to fructose intake, which will be useful for creating preventive campaigns aimed at promoting a healthy lifestyle. This includes changing dietary habits to encourage a healthy diet and reducing obesity in the population.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents of both sexes aged 3-6 years and 12-16 years, as interest groups for the assessment of hepatic steatosis induced by fructose consumption.
* Children with overweight (defined by BMI > 97 year old percentile for children under 5 years old; and BMI >85 year old percentile for children over 5 years old) or obesity (defined by BMI > 99 percentile for children under 5 years of age; and BMI > 97 percentile for children over 5 years of age)

Exclusion Criteria:

* Children and adolescents not in that age group:
* Children and adolescents with different liver diseases of NAFLD, as it is the interest of the study
* Children and adolescents with genetic obesity or secondary obesity since the interest of the study is obesity caused by excessive calorie intake
* Children and adolescents included in diet-therapy regimen with different dietary styles from the Mediterranean or Western diet (example ketogenic diet, FoadMap (fermentable oligosaccharides, disaccharides, monosaccharides and polyols) diet, vegan/vegetarian diet) to avoid bias in the interpretation of the microbial signature (the microbial signature of the Western and Mediterranean diet is known in the literature);

Ages: 3 Years to 16 Years | Sex: All
Age Groups: Child
Study Population: 100 pediatric patients with overweight and obesity
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2025-03-05 (Estimated); Study Completion 2026-03-02 (Estimated)

PRIMARY OUTCOMES:
assessment of fructose intake with questionnaires | evaluation of fructose intake through study completion, an average of 1 year
  assessment of fructose intake in preschool children and adolescent with obesity or overweight, using questionnaires with multiple answers
correlation of fructose consumption with hepatic complications, detected trough echo-abdomen and blood analysis | assessment of fructose intake in correlation with hepatic complications through study completion, an average of 1 year
  assessment of fructose intake in correlation with hepatic complications using echo-abdomen and blood analysis as detection methods
Correlation of fructose consumption with bone metabolism, detected through QUS | assessment of fructose intake in correlation with bone metabolism through study completion, an average of 1 year
  assessment of fructose intake in correlation with bone metabolism, using QUS as detection method

SECONDARY OUTCOMES:
Characterization of the concentration of intestinal microorganisms | Evaluation of microbiota after 12 months
  Characterization of microorganisms present in the gastrointestinal tract and their microbial activity
Evaluate sociodemographic and cultural determinants with questionnaires ( questions with multiple answers) | Evaluation of sociodemographic data after 12 months
  Evaluate sociodemographic and cultural determinants, and differences between Northern and Southern Italy through the use of questionnaires. Assessment scales will not be used, but will be a collection of data evaluated in a descriptive manner. There are no maximum and minimum, but what we will get from the questionnaires will be a descriptive overview of the population in Italy.

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Prodam, MD PHD, Principal Investigator — AOU Maggiore della Carità
Locations (1):
- SCDU Pediatria, AOU Ospedale Maggiore della Carità, Novara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marriott BP, Cole N, Lee E. National estimates of dietary fructose intake increased from 1977 to 2004 in the United States. J Nutr. 2009 Jun;139(6):1228S-1235S. doi: 10.3945/jn.108.098277. Epub 2009 Apr 29. PMID 19403716
- [Background] Alisi A, Carpino G, Nobili V. Paediatric nonalcoholic fatty liver disease. Curr Opin Gastroenterol. 2013 May;29(3):279-84. doi: 10.1097/MOG.0b013e32835ff95e. PMID 23493072
- [Background] Zhang DM, Jiao RQ, Kong LD. High Dietary Fructose: Direct or Indirect Dangerous Factors Disturbing Tissue and Organ Functions. Nutrients. 2017 Mar 29;9(4):335. doi: 10.3390/nu9040335. PMID 28353649
- [Background] Lanaspa MA, Sanchez-Lozada LG, Cicerchi C, Li N, Roncal-Jimenez CA, Ishimoto T, Le M, Garcia GE, Thomas JB, Rivard CJ, Andres-Hernando A, Hunter B, Schreiner G, Rodriguez-Iturbe B, Sautin YY, Johnson RJ. Uric acid stimulates fructokinase and accelerates fructose metabolism in the development of fatty liver. PLoS One. 2012;7(10):e47948. doi: 10.1371/journal.pone.0047948. Epub 2012 Oct 24. PMID 23112875
- [Background] Hostmark AT, Sogaard AJ, Alvaer K, Meyer HE. The oslo health study: a dietary index estimating frequent intake of soft drinks and rare intake of fruit and vegetables is negatively associated with bone mineral density. J Osteoporos. 2011;2011:102686. doi: 10.4061/2011/102686. Epub 2011 Jul 2. PMID 21772969
- [Background] WHO Multicentre Growth Reference Study Group. WHO Child Growth Standards based on length/height, weight and age. Acta Paediatr Suppl. 2006 Apr;450:76-85. doi: 10.1111/j.1651-2227.2006.tb02378.x. PMID 16817681
- [Background] Huybrechts I, Bornhorst C, Pala V, Moreno LA, Barba G, Lissner L, Fraterman A, Veidebaum T, Hebestreit A, Sieri S, Ottevaere C, Tornaritis M, Molnar D, Ahrens W, De Henauw S; IDEFICS Consortium. Evaluation of the Children's Eating Habits Questionnaire used in the IDEFICS study by relating urinary calcium and potassium to milk consumption frequencies among European children. Int J Obes (Lond). 2011 Apr;35 Suppl 1:S69-78. doi: 10.1038/ijo.2011.37. PMID 21483425
- [Background] Cavicchia PP, Steck SE, Hurley TG, Hussey JR, Ma Y, Ockene IS, Hebert JR. A new dietary inflammatory index predicts interval changes in serum high-sensitivity C-reactive protein. J Nutr. 2009 Dec;139(12):2365-72. doi: 10.3945/jn.109.114025. Epub 2009 Oct 28. PMID 19864399
- [Background] Takahashi Y, Fukusato T. Histopathology of nonalcoholic fatty liver disease/nonalcoholic steatohepatitis. World J Gastroenterol. 2014 Nov 14;20(42):15539-48. doi: 10.3748/wjg.v20.i42.15539. PMID 25400438
- [Background] Nier A, Brandt A, Conzelmann IB, Ozel Y, Bergheim I. Non-Alcoholic Fatty Liver Disease in Overweight Children: Role of Fructose Intake and Dietary Pattern. Nutrients. 2018 Sep 19;10(9):1329. doi: 10.3390/nu10091329. PMID 30235828
- [Background] Anderson EL, Howe LD, Jones HE, Higgins JP, Lawlor DA, Fraser A. The Prevalence of Non-Alcoholic Fatty Liver Disease in Children and Adolescents: A Systematic Review and Meta-Analysis. PLoS One. 2015 Oct 29;10(10):e0140908. doi: 10.1371/journal.pone.0140908. eCollection 2015. PMID 26512983

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-21): https://cdn.clinicaltrials.gov/large-docs/67/NCT06365567/Prot_SAP_000.pdf